CLINICAL TRIAL: NCT06970145
Title: Safety and Efficacy of Anlotinib in the Treatment of Recurrent Craniopharyngioma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-156
Record Dates: First submitted 2025-04-22; First posted 2025-05-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Craniopharyngiomas
Keywords: Anlotinib; Craniopharyngiomas; Targeted therapy
MeSH Terms: conditions — Craniopharyngioma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-center, open-label, single-arm, experimental clinical trial without any control group (Experimental): This is a single-center, open-label, single-arm, experimental clinical trial without any control group. The study was conducted in patients with recurrent craniopharyngiomas
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib Hydrochloride Capsules (12mg),Chiatai Tianqing Pharma (China).
  Other Names: Anlotinib Hydrochloride Capsules

SUMMARY:
Primary Aim:

To assess the objective remission rate (ORR) of patients with recurrent craniopharyngiomas treated with anlotinib .

Secondary Aims:

1. To assess progression-free survival (PFS) and overall survival (OS) of patients with recurrent craniopharyngiomas treated with anlotinib.
2. To analyze the disease control rate (DCR) of the anlotinib treatment regimen in patients with recurrent craniopharyngiomas, including the proportion of patients in complete remission, partial remission and stable disease.
3. Monitor and evaluate the safety of anlotinib, especially the occurrence of drug-related adverse events (AEs) .

DETAILED DESCRIPTION:
This study is a single-center, open-label, single-arm clinical trial designed to evaluate the safety and efficacy of anlotinib in the treatment of recurrent craniopharyngioma. Primary endpoints include progression-free survival (PFS), overall survival (OS), and objective remission rate (ORR), with assessment of treatment-related adverse events and quality of life.

Analysis Set:

Full Analysis Set (FAS): includes all patients who are randomized into the study, have received at least received at least one dose of study drug and have measurable baseline tumors.FAS will be used for efficacy FAS will be used for efficacy analysis. Per-Protocol Set (PPS): In the FAS, patients with at least one post-dose tumor imaging evaluation and a compliant tumor.

PPS: In the FAS, patients with at least one post-dose tumor imaging assessment, good compliance, and no significant violations or deviations from the trial protocol.

PPS will be used for secondary efficacy analysis. Safety Set (SS): Includes all patients who have received at least one dose of drug therapy and have completed at least one safety assessment.

SS will be used for safety analysis.

Sample size determination:

This is an experimental clinical study with the primary objective of assessing the safety and preliminary efficacy of the drug.

The sample size was designed to be relatively small due to resource constraints and the nature of experimental clinical studies. Based on the literature references and study design, we expected to enroll approximately 57 subjects.

Statistical analysis All statistical analyses will be performed using SAS 9.2 statistical analysis software. Separate independent efficacy and safety analyses will be performed, and no control will be established.

efficacy and safety analyses will be performed separately, with no control group and no between-group comparisons.ORR and DCR will be described using frequency and percentage, PFS and OS will be described using frequency and percentage.

ORR and DCR were described using frequency and percentage, PFS and OS were estimated by Kaplan-Meier method for survival, and All treatment-related adverse events were recorded and analyzed according to CTCAE 5.0 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, regardless of gender
2. recurrent craniopharyngioma (recurrence after total resection or regrowth of residual tumor) confirmed by pathology and imaging data
3. predominantly cystic or solid recurrence of the tumor
4. measurable lesions (according to the RECIST criteria)
5. Karnofsky score ≥ 70, expected survival ≥ 3 months
6. laboratory parameters (liver and kidney function, blood tests, etc.) within the normal range or under control
7. signed informed consent and willing to participate in the study

Exclusion Criteria:

1. Have a combination of other intracranial tumors or severe brain lesions
2. primary craniopharyngioma
3. have severe uncontrolled heart, lung, kidney, or liver disease
4. children, pregnant or breastfeeding women
5. prior treatment with the same investigational drug
6. active infections, including HIV, HBV, or HCV infections
7. patients who do not meet the contraindications to the medication
8. have a history of severe allergy to the investigational drug
9. have psychiatric illnesses or cognitive impairments and unable to complete follow-up visits or understand the purpose of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of tumor volume on imaging (MRI) | Through study completion, an average of 1 year
  Measurement of tumor volume on imaging (MRI): A*B*C/2 (A,B,C are the maximum length, width, and height of the tumor, respectively)

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Nanfang Hospital, Department of Neurosurgery, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No